CLINICAL TRIAL: NCT00494845
Title: Mindfulness Meditation for Chronic Low Back Pain in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Natalia Morone, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PRO07020074; UL1RR024153 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2016-01

CONDITIONS: Low Back Pain
Keywords: Mindfulness; Elderly; Chronic Illness; Back Pain; Chronic Low Back Pain; Older adults over the age of sixty-five; MMSE score of over 23; Speaks English
MeSH Terms: conditions — Low Back Pain; Chronic Disease; Back Pain | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 8-week Mindfulness Program for chronic low back pain
  Interventions: Behavioral: Mindfulness
- Comparison (Active Comparator): 8-week health education program
  Interventions: Behavioral: Control: Health Education Class

INTERVENTIONS:
Behavioral: Mindfulness — 8-week mindfulness program will be compared to an education control group.
  Arms: Intervention
Behavioral: Control: Health Education Class — 8-week education program
  Arms: Comparison

SUMMARY:
Among mind-body therapies, there is evidence for an association between pain reduction and mindfulness meditation. Mindfulness meditation provides a potentially safe, effective, nonpharmacologic, noninvasive, simple method for pain relief and increased function that could be used for the frailest older adult. Additionally, mindfulness meditation addresses the multiple dimensions that are affected by chronic pain. The primary objective of this study is to determine the impact of an 8-week mindfulness-based stress reduction program on physical function and pain severity in community dwelling older adults with chronic low back pain. Using a randomized controlled experimental design, 80 community dwelling older adults ≥ age 65 with chronic low back pain will receive either (1) the MBSR program, or (2) an 8-week education program. Prior to initiating the program, immediately after the last program session, and 6 months later, the following parameters will be assessed: (1) pain severity, (2) disability/physical function, (3) objectively measured physical performance, (4) psychosocial function (including mood, self-efficacy, self-rated health, coping, stress, quality of life (QOL), mindfulness and pain-related fear), (5) sleep, (6) pain-related appetite reduction and, (7) time and frequency of meditation. All measures are self-report except for the physical performance measure.

DETAILED DESCRIPTION:
3.0 Research Design and Methods This pilot experimental study is designed as a randomized, education controlled clinical trial of mindfulness meditation for CLBP. A sample of 80 older adults 65 years of age and older will be recruited from a chronic pain clinic, general medicine research registry, posted flyers, and newspaper advertisements over an 18-month period. Eligibility will be determined by self-report from a checklist reviewed with potential participants over the phone. Pre-intervention study participants will be consented and study measures obtained. After consent and baseline measures, participants will be randomized using a simple randomization process with no stratification using a software generated randomization plan. After randomization, participants in the intervention group will receive the intervention of eight weekly 90-minute mindfulness meditation sessions. Controls will receive an 8-week health education program. Subject evaluation and each program will occur at the University of Pittsburgh Center for Research on Health Care (CRHC) which has subject examination areas as well as a classroom and a nearby parking structure. Subjects will be assessed weekly over the telephone during the intervention or health education program with a subset of measures administered at baseline. Immediately post-intervention or education program the complete set of measures will be administered again to participants and controls. Subjects will be assessed monthly by telephone for five months after completion of the MBSR or health education program with the same subset of baseline measures. Six months after the intervention is completed, participants will be asked to return to the CRHC and complete the entire set of measures a third time and any mindfulness meditation the intervention group continues to do at home will be quantified.

3.2 Procedures

3.2.2 Entry Phase: All 40 subjects who are included based upon the screening criteria will receive identical pre-treatment baseline assessments. Data will be collected and interviewer-administered by a trained research assistant at the University of Pittsburgh CRHC.

After successful telephone screening, written informed consent, and baseline examination, all eligible research subjects entering this study will be randomized into one of two treatment groups; 1) education group (control) or 2) mindfulness meditation (treatment). The randomization process will be performed using statistical software with a random-number generator to generate a randomization list before the study commences.

3.2.4 Intervention Phase: Participants will be seen in a group format once a week for 90 minutes for 8-weeks. All sessions will be led by a facilitator experienced in teaching the MBSR program and who has undergone teacher training in at least one intensive (≥ 50 hours) MBSR teacher training program conducted by the University of Massachusetts Medical School Center for Mindfulness prior to the intervention. All sessions will occur at the University of Pittsburgh Center for Research on Health Care (CRHC).

MBSR Intervention: The intervention is based on the work of Jon Kabat-Zinn at the Massachusetts Medical Center. He has adapted Eastern methods of mindfulness meditation to a Western audience. Three techniques of mindfulness meditation will be taught. These techniques take regular activities like sitting, walking and lying down and transform them into a meditation through directed breathing and mindful awareness of thoughts and sensations.

The techniques used are: 1) the body scan, where in a lying position, the participant is guided to place their attention non-judgmentally on each area of the body from the toes to the top of the head and directing the breath to each region in turn, 2) sitting practice, which is focused attention on breathing while sitting on a chair or cross-legged on the floor, 3) walking meditation, which is mindful slow walking with focused attention on body sensation and /or breathing (15).

During the first week participants will be introduced to the principles and practice of mindfulness meditation. The homework requirement of daily meditation (six of seven days/week) lasting 50 minutes (45 minutes of meditation, 5 minutes to complete a log) will be reviewed. Support materials of audiotape or CD recording, daily log and reading materials will be handed out. The audiotape or CD recording is a 45 minute recording of the steps in the body scan meditation and a 30 minute recording of the sitting meditation that guides participants in meditation. The reading materials will be reviewed during the sessions and are not part of the homework. The log is described later in this protocol. The body scan technique will be taught at the first session. The group will meditate together using the body scan technique for 45 minutes at the first and most subsequent sessions. If physical discomfort should arise during any meditation participants will be encouraged to change to a more comfortable position. There is not a minimum amount of time required to stay in one position.

During the second and following weeks the sessions will include a general discussion of the participants' experience with the meditation method, including problem solving regarding obstacles to the meditation practice. Theoretical material related to meditation, relaxation, pain and the mind/body connection will be presented at this time. About 30 minutes will be spent at each session in these discussions. Also during the second week, quiet sitting meditation will be introduced. The group will practice together using the sitting meditation technique for 15 minutes during this and at the beginning of subsequent sessions.

At the fifth week's session, walking meditation will be introduced. Therefore, the structure of each session will be one hour (total) of meditation and 30 minutes of discussion.

Health Education Control Program: A convincing comparison group is essential for subject recruitment and retention as well as essential for controlling for key components of the MBSR program. Therefore, we will create a comparison group that will control for time, group size and facilitator time. We are basing the 8-week health education program on a successful aging curriculum that has been used in other trials (80, 81). The health education curriculum will involve lectures, group interaction and homework assignments based on the health topics discussed. Sessions will include topics such as (a) medications, (b) foot care, (c) traveling, and (d) nutrition. Additionally, subjects will be given materials to promote participation and retention in the program. For example, participants will receive the "passport" to health, available from the Pennsylvania Department of Aging. It is a small booklet that seniors fill out with essential health information such as medical problems and medications. Filling out the passport will be one of the homework assignments. The health education group will receive ongoing staff attention. This person will coordinate and be present at all classes. The consistent presence of a class coordinator will control for the facilitator contact of the MBSR program. This type of intervention is deemed scientifically "inert" (i.e., not affecting the outcomes of interest in this trial). Previous trials such as the LIFE-P trial demonstrated an excellent retention rate of 91.5% (82).

3.3 Data Collection and Statistical Considerations

3.3.1 Outcome measures: Outcome measures were chosen to reflect our primary aim of determining the impact of the MBSR program on physical function and pain. To reflect our secondary aim of determining the impact of the MBSR program on the multidimensional aspects of chronic pain, comprehensive psychosocial, sleep and appetite measures were decided on. Outcome measures were also chosen because of their demonstrated feasibility, reliability, and validity in older adults with chronic pain.

Questionnaires will be administered at baseline, completion of the 8-week program, and 6-month follow up include 1) measures of physical ability with the SF-36 Physical Function Scale (49) , Roland and Morris Disability Questionnaire (51), Short Physical Performance Battery (52, 53); 2) measure of pain with the McGill Pain Questionnaire (MPQ), Short Form (54) and The Pain Thermometer (51); 3) measures of psychosocial function with the SF-36 Health Survey (55), Geriatric Depression Scale (57), Chronic Pain Acceptance Questionnaire (58), Multidimensional Pain Inventory (60), Catastrophizing Scale of the Cognitive Strategies Questionnaire (61), Fear-Avoidance Beliefs Questionnaire (62), Chronic Pain Self-Efficacy Scale (65), Self-rated heath (SRH) using standardized methods (66, 67); 4) measures of mindfulness with the Kentucky Inventory of Mindfulness Skills (68) and Mindful Attention Awareness Scale (MAAS) (69, 70); 5) measures of stress with the well-validated Perceived Stress Scale (71); 6) measures of sleep with a modified Pittsburgh Sleep Quality Index (73); 7) measures of appetite by evaluating pain-related appetite impairment.

3.3.2 Evaluation of Treatment Outcome:

Weekly Assessments: To examine the process of change, brief (15 minutes) weekly telephone evaluations of major important domains (pain, physical function, psychosocial function, sleep) will be conducted. The measures are a subset of the collected baseline measures (see D.3.3.1). These data will allow a detailed examination of the temporal association of the individual weeks of the 8-week MBSR program with the primary outcomes of pain and physical function as well as secondary outcomes of psychosocial function. It will also allow a detailed examination of the temporal relationship between time and frequency meditating and the primary and secondary outcomes. All measures will be collected weekly over the telephone one-two days before the treatment sessions. These measures will be collected by the research assistant who will be blinded to randomization assignment. These weekly dependent measures will include assessment of pain, physical function, psychosocial function and sleep with 1) the SF-36 Physical Function scale, 2) self-reported pain in the past week on a scale of 0-100, 3) the short-form of the Multidimensional Pain Inventory, 4) subjects' reports of any pain medication usage (including OTC) during the previous week (type, dosage, and frequency), tracked with diaries, 5) the five item MAAS, 6) the Pittsburgh Sleep Quality Index; and 7) Acute Illness/injury or exacerbation of comorbidity will be assessed with yes/no questions and if answered positively, the participant will be asked to describe the event.

Post-program Evaluation: Within one week of completing the 8-week MBSR or health education program, subjects will return to the CRHC and will be evaluated in a manner similar to the preprogram evaluation. That is, all measures outlined in D.3.3.1 will be repeated. Independent global ratings of improvement on a 5 point scale also will be made by the research subjects (83).

Six-month follow up (FU): Subjects will be interviewed by telephone at monthly intervals after the post-program evaluation for 5 months. Brief structured interviews will assess subjects' perceptions of improvement since treatment, time and frequency of meditation for the treatment group, current pain intensity, physical function, mindfulness and sleep (using the same measures collected weekly). In addition, medication use and additional treatment seeking will be assessed. At 6 months post-treatment, subjects will be asked to return to the CRHC for an evaluation that will be identical to the pre- and post-treatment evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Have intact cognition (Mini-Mental Status Exam (MMSE) >23)
* CLBP, defined as moderate pain occurring daily or almost every day for at least the previous three months
* Speak English.

Exclusion Criteria:

* Do not meet the above inclusion criteria
* Have previously participated in a mindfulness meditation program
* Have serious underlying illness (like malignancy, infection, unexplained fever, weight loss or recent trauma) causing their pain,
* Are non-ambulatory, or have severely impaired mobility (i.e., require the use of a walker): since measurement of physical performance in the proposed study includes timed chair rise, gait velocity, and standing balance, conditions other than back pain that could negatively impact these measures may confound our study results
* Severe visual or hearing impairment: since this study will involve questionnaires and telephone evaluations, severe visual and/or hearing impairments may interfere with data collection
* Significant pain in parts of the body other than the lower back or acute back pain: since we will be specifically evaluating chronic low back pain, we do not want to confound the outcome data with pain from other areas or with acute pain. Thus only subjects with chronic back pain severity that is greater than pain severity elsewhere in the body will be included
* Acute or terminal illness: To insure weekly participation and a six month follow-up, subjects with an acute or terminal illness will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Determine the impact of an 8-week mindfulness-based stress reduction program on physical function and pain severity in community dwelling older adults with chronic low back pain. | One year
Determine the impact of an 8-week mindfulness-based stress reduction program on psychosocial function, sleep, and appetite in older adults with chronic low back pain. | One year
Determine the impact of time and frequency of mindfulness meditation on physical function and pain severity. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morone, MD, MS, Principal Investigator — University of Pittsburgh